CLINICAL TRIAL: NCT01366703
Title: Optimized Heart Failure Therapy Through Continuous Monitoring. The PHARAO Multi-centre Study
Brief Title: Optimized Heart Failure Therapy Through Continuous Monitoring
Acronym: pharao
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kennemer Gasthuis (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. R. Tukkie MD PhD FESC, Dr., Kennemer Gasthuis
Other Study IDs: pharao multicentre study
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure
Keywords: heart failure; implantable loop recorder
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- heart failure patients: stable heart failure patients, NYHA 1-2, EF > 35%, no AF, No OAC, CHADS score >2
  Interventions: Device: implantable loop recorder Medtronic reveal XT Full view

INTERVENTIONS:
Device: implantable loop recorder Medtronic reveal XT Full view — Medtronic Reveal implantable loop recorder with home-monitoring using carelink will be implanted in every patient and used to continuously monitor the patients during follow-up to detect symptomatic and asymptomatic arrythmias during follow-up
  Other Names: Medtronic reveal XT Full view

SUMMARY:
Patients with heart failure have a high incidence of atrial fibrillation (AF)and re-admission for heart failure. New methods have been developed to continuously monitor arrhythmia's and heart failure parameters. One such method is implantation of an implantable loop recorder. Also home-monitoring is available for continuous monitoring and information sending to the treating physicians, with improving detection of atrial fibrillation (AF) and/or other sever arrhythmia's we hope to improve patient care.

Objective of the study:

To investigate the clinical efficacy in detecting clinically relevant arrhythmia's (especially AF) of the Reveal XT in patients with mild to moderate heart failure and elevated risk factor for stroke and transient ischemic attack (TIA)(CHADS-score >2), currently not treated with oral anticoagulation (OAC).

Study design:

In 50 stable sinus rhythm (no known AF)patients with New York health Association (NYHA class) 2-3, a CHADS2-score>2 and no indication for a implantable cardioverter-defibrillator (ICD) or pacemaker (PM) or OAC. Patients are put on home-monitoring (CareLink) and regular outward clinic visits. The number of relevant arrhythmia's detected will count for the primary endpoint. Also the number of medication changes and institution of OAC.

Study population:

50 stable patients, recruited from the outward clinic. NYHA class 2-3. Reveal XT implantation. CHADS2-score 2 or more. No indication for ICD/PM or OAC. No AF known.

Primary study parameters/outcome of the study:

Primary endpoints

* AF burden and AF episodes detected
* Detected other relevant arrhythmia's like SVT's (not AF) or ventricular tachycardias (VT's) or bradycardias
* % patients on OAC after 1 year follow-up
* Number of clinically relevant patient activated events
* Number of treatment policy changes based on the Reveal XT

Secondary study parameters/outcome of the study

* specificity of AF detection algorithm by the Reveal
* Predictive value of the cardiac Compass data to predict worsening heart failure episodes.

DETAILED DESCRIPTION:
no additional description needed

ELIGIBILITY:
Inclusion Criteria:

* EF > 35%
* NYHA 2-3
* No AF documented
* Not on OAC

Exclusion Criteria:

* use of OAC
* documented AF > 30 sec
* planned or actual PM/ICD
* life-expectancy < 1 year
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with stable heart failure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
registered arrhythmias with implantable loop recorder during follow-up period | 1 year follow-up after last included patient
  Primary study parameters/outcome of the study:
  * AF burden en AF episodes detected
  * Detected other relevant arrhythmia's like supraventricular tachycardia's (SVT's, not AF) or ventricular tachycardia's (VT's) or bradycardias
  * % patiënts on OAC after 1 year follow-up
  * Number of clinically relevant patient activated events
  * Number of treatment policy changes based on the Reveal XT

SECONDARY OUTCOMES:
prediction of worsening heart failure through cardiac compass | during follow-up (1 year after last included patient)
  Predective value of the cardiac Compass data to predict worsening heart failure episodes.

CONTACTS AND LOCATIONS:
Overall Officials: raymond tukkie, MD PhD, Principal Investigator — Kennemer Gasthuis
Locations (5):
- Netherlands (5):
  - Rijnstate ziekenhuis, Arnhem
  - Deventer Ziekenhuis, Deventer
  - Martini Ziekenhuis, Groningen
  - Kennemer gasthuis, Haarlem
  - Rijnland Ziekenhuis, Leiderdorp